CLINICAL TRIAL: NCT01408563
Title: A Phase II Study of Reduced Intensity Double Umbilical Cord Blood Transplantation Using Fludarabine, Melphalan, and Low Dose Total Body Radiation
Brief Title: Reduced Intensity Double Umbilical Cord Blood Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Zachariah Michael DeFilipp, Hematology/Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-085
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-12

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Multiple Myeloma; Chronic Lymphocytic Leukemia; Acute Myelogenous Leukemia
Keywords: NHL; lymphoma; leukemia; myelodysplastic disorder; aplastic anemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Lymphoma; Leukemia; Anemia, Aplastic | interventions — fludarabine; fludarabine phosphate; Melphalan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine/Melphalan/TBI (Experimental): All patients receive same therapy
  Interventions: Drug: Fludarabine; Drug: Melphalan; Radiation: Total Body Radiation; Biological: Cord Blood

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m2/day IV x 6 days
  Other Names: Fludara
Drug: Melphalan — 100 mg/m2/day IV x 1 day
Radiation: Total Body Radiation — 200 cGy on Day 0
Biological: Cord Blood — 2 cord blood units IV

SUMMARY:
This trial will use two cord blood units for transplantation using a reduced intensity regimen rather than using intense doses of chemotherapy and radiation therapy. Two cord blood units (double cord blood) are being used, as the numbers of blood cells in one unit are too few to allow successful growth of these cells.

Because the risk of infection, particularly virus infection, is high after double cord blood transplant, this study seeks to reduce the rise of virus infection by using a reduced intensity regimen without a medicine called antithymocyte globulin (ATG), as used in prior cord blood transplants. Subjects will receive two chemotherapy drugs, melphalan and fludarabine, and low dose of total body radiation (one treatment) instead of the ATG. The number of patients with virus infections in this study will be compared to our prior experience using the ATG.

DETAILED DESCRIPTION:
Subjects will receive their transplants as in-patients.

* IV-Catheter

  * one or two IV catheters will be placed on the day of hospital admission
* Conditioning

  * Fludarabine IV six days before transplant (days -7, -6, -5. -4, -3, -2)
  * Melphalan IV (day -1)
  * Total body radiation on day 0 (same day as transplant)
* Immunosuppressive Therapy

  * Tacrolimus and sirolimus beginning day -3, daily for 6-9 months post-transplant. Given IV as in-patient, orally as out-patient
* Infusion of Cord Blood units

  * 2 cord blood units IV on Day 0 Routine post-transplant supportive care will be provided

ELIGIBILITY:
Inclusion Criteria:

* Hematologic malignancy for whom allogeneic stem cell transplantation is deemed clinically appropriate
* Appropriate candidate for reduced intensity regimen, according to the treating physician
* Lack of 6/6/ or 5/6 HLA-matched related, 8/8/ HLA-matched unrelated donor, or unrelated donor not available with a time frame necessary to perform a potentially curative stem cell transplant
* Able to comply with the requirements for care after allogeneic stem cell transplantation

Exclusion Criteria:

* Cardiac disease: symptomatic congestive heart failure or evidence of left ventricular dysfunction
* Pulmonary disease: symptomatic chronic obstructive lung disease, symptomatic restrictive lung disease
* Renal disease
* Hepatic disease
* Neurologic disease: symptomatic leukoencephalopathy, active CNS malignancy or other neuropsychiatric abnormalities believed to preclude transplantation
* HIV-positive
* Uncontrolled infection
* Pregnant or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachariah DeFilipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fludarabine/Melphalan/TBI
Started | 33
Received Transplant | 31
Completed | 31
Not Completed | 2
Not completed — Ineligible after consent/ registration | 2

BASELINE CHARACTERISTICS:
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis.
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 57 [21 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31
Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status:
  * 0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  * 1 - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  * 2 - Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  Participants
    0 | 10
    1 | 19
    2 | 2
Disease [Count of Participants; unit: Participants]
  Acute Lymphoblastic Leukemia (ALL) | 2
  Acute Myeloid Leukemia (AML) | 11
  Hodgkin's Disease (HD) | 1
  Myelodysplastic Syndromes (MDS) | 8
  Myeloproliferative Disorder (MPD) | 2
  Non-Hodgkin Lymphoma (NHL) | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinically Significant Infection
Description: The one year significant infection rate (infections requiring medical intervention) after double umbilical cord blood transplant using a novel conditioning regimen of fludarabine/melphalan/low dose total body radiation. The data is shown as the number of significant infections participants experienced during the first year, measured from the start of treatment.
Time Frame: 1 Year
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
Participants
  0 Infections | 12
  1 Infection | 14
  2 Infections | 5

2. Secondary Outcome: Median Time to Neutrophil Engraftment
Description: The median number of days measured from the time of transplantation, until the first documented neutrophil engraftment. neutrophil engraftment is defined as the first of 3 consecutive days of absolute neutrophil count > 500 neutrophils per microliter of blood.
Time Frame: From the time of transplantation, until the time of neutrophil engraftment, median duration of 24 days
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis. In addition to those two participants, the 8 participants that did not achieve engraftment were not included in the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 23
Days | 24 [1 to 54]

3. Secondary Outcome: Median Time to Platelet Engraftment
Description: The time to platelet engraftment is measured from the time of transplantation until the time of first documented platelet engraftment. Platelet engraftment is defined as a platelet count ≥ 20,000/µL for three consecutive measurements over three or more days. The first of the three days will be designated the day of platelet engraftment. Subjects must not have had platelet transfusions during the preceding 3 days or in the following 7 days after the day of engraftment, unless the platelet transfusion is being given specifically to achieve a platelet threshold to allow an elective invasive procedure, such as a central catheter removal.
Time Frame: From the time of transplantation, until the time of platelet engraftment, median duration of 52 days
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis. In addition to those two participants, the 10 participants that did not achieve engraftment were not included in the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 21
Days | 52 [21 to 89]

4. Secondary Outcome: Number of Participants With Primary Graft Failure
Description: Primary graft failure is defined as the failure to achieve an absolute neutrophil count (ANC) >500/ µL by day 42, in the absence of relapse.
Time Frame: From the time of transplantation until 42 days post transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
Participants | 8

5. Secondary Outcome: Rates of Grade II-IV and Grade III-IV Acute Graft Versus Host Disease (GVHD) at 100 Days
Description: Acute GVHD is assessed using Consensus Criteria:
  Organ Classifications:
  * 0: No rash due to GVHD; Bilirubin < 2 mg/dL; < 500 mL diarrhea/ day
  * 1: Maculopapular rash < 25% of body surface; Bilirubin 2-3 mg/dL; 500 to 999 mL diarrhea/ day or persistent nausea with histologic evidence of GVHD in stomach/ duodenum
  * 2: Maculopapular rash 25-50% of body surface; Bilirubin 3.1-6 mg/dL; 1,000 to 1,499 mL diarrhea/ day
  * 3: Maculopapular rash > 50% of body surface; Bilirubin 6.1-15 mg/dL; 1,500 or more mL diarrhea/ day
  * 4: Generalized erythroderma with bullous formation; Bilirubin > 15 mg/dL; Severe abdominal pain with or without ileus
  Overall Clinical Grade:
  * 0: No Stage 1-4 of any organ
  * I: Stage 1-2 rash and no liver or gut involvement
  * II: Stage 3 rash, or Stage 1 liver involvement, or Stage 1 gut involvement
  * III: None to Stage 3 skin rash with Stage 2-3 liver involvement, or Stage 2-4 gut involvement
  * IV: Stage 4 skin rash, or Stage 4 liver involvement
Time Frame: 100 Days
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
percentage of participants | 16 [5.7 to 31]

6. Secondary Outcome: The Rate of Chronic GVHD
Description: Chronic Graft Versus Host Disease (GVHD) is assessed using the National Institutes of Health (NIH) consensus criteria.
Time Frame: From the time of transplantation until the time of chronic GVHD onset, up to 1 year
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
percentage of participants | 21 [8.1 to 37]

7. Secondary Outcome: 100-day Treatment Related Mortality
Description: The percentage of treatment related participant deaths within 100 days of receiving umbilical cord blood transplantation. All deaths in the absence of relapse of the primary malignancy will be considered treatment related mortality.
Time Frame: 100 Days
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
percentage of participants | 9.7 [2.4 to 23]

8. Secondary Outcome: Immune Reconstitution - Median CD4 Count at 12 Months
Time Frame: 1 Year
Population: CD4 counts were only available for 11 participants at the 12 months time point
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 11
cells/mm3 | 362.4 [125.3 to 1157.8]

9. Secondary Outcome: Relapse-free Survival
Description: The percentage of participants that have not died or had disease progression by two years. Relapse is defined by either morphological or cytogenetic evidence of the original malignancy consistent with pre-transplant features.
Time Frame: 2 years
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
percentage of participants | 49 [30 to 66]

10. Secondary Outcome: Overall Survival
Description: The percentage of participants alive at two years
Time Frame: 2 years
Population: The two participants found to be ineligible after being consented and registered were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
percentage of participants | 55 [35 to 71]

11. Secondary Outcome: 1 Year Relapse Rate
Description: The percentage of participants that relapsed within 12 months. Relapse is defined by either morphological or cytogenetic evidence of the original malignancy consistent with pre-transplant features.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
percentage | 20 [4 to 27.3]

12. Secondary Outcome: Rate of Post-transplant Lymphoma
Description: The number of participants that were found to have lymphoma post-transplant.
Time Frame: 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
Participants | 0

13. Secondary Outcome: Median Thrombopoietin Levels After Transplant
Time Frame: 30 Days
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Fludarabine/Melphalan/TBI
Number analyzed (Participants) | 31
pg/mL | 2500 [320 to 4000]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed from the start of treatment until the end of follow-up, up to two years.
Description: The two participants found to be ineligible after being consented and registered were excluded from the analysis.
Arm/Group | Fludarabine/Melphalan/TBI
All-Cause Mortality (participants affected / at risk) | 1/31
Serious Adverse Events (participants affected / at risk) | 10/31
Other Adverse Events (participants affected / at risk) | 26/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine/Melphalan/TBI (N=31)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine/Melphalan/TBI (N=31)
Abdominal pain (Gastrointestinal disorders) | 4 (11)
Acidosis (Metabolism and nutrition disorders) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 3 (8)
Anorexia (Metabolism and nutrition disorders) | 4 (7)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 6 (21)
Blood bilirubin increased (Investigations) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 12 (15)
Encephalitis infection (Infections and infestations) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (9)
Fever (General disorders) | 4 (6)
Headache (Nervous system disorders) | 7 (17)
Hypertension (Vascular disorders) | 4 (12)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung infection (Infections and infestations) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 7 (14)
Nausea (Gastrointestinal disorders) | 9 (18)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 6 (16)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT01408563/Prot_SAP_000.pdf